CLINICAL TRIAL: NCT06973096
Title: Phase 1 Open-label Study Evaluating the Safety of CART-EGFR-IL13Rα2 Cells in Patients With Newly Diagnosed, EGFR-Amplified, MGMT-unmethylated Glioblastoma Following Completion of Initial Radiotherapy
Brief Title: CART-EGFR-IL13Ra2 in Newly Diagnosed GBM Following Initial Radiotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 03325
Record Dates: First submitted 2025-05-01; First posted 2025-05-15 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Level 1 (Experimental): Dose Level 1 (DL1): will receive single fixed dose of 2.5x10^7 CART-EGFR-IL13Ra2 cells via intracerebroventricular (ICV) injection on Day 0.
  Interventions: Drug: CART-EGFR-IL13Ra2 cells
- Dose Level -1 (DL-1) (Experimental): Dose Level-1 (DL-1): will receive single fixed dose of 1x10^7 CART-EGFR-IL13Ra2 cells via intracerebroventricular (ICV) injection on Day 0.
  This dose level will only be explored if there are at least two TLTs observed at DL1.
  Interventions: Drug: CART-EGFR-IL13Ra2 cells

INTERVENTIONS:
Drug: CART-EGFR-IL13Ra2 cells — autologous T cells transduced with a bicistronic lentiviral vector containing a murine scFv targeting EGFR epitope 806 and a humanized scFv targeting IL13Ra2; both scFvs are fused to the 4-1BB and CD3ζ signaling domains.

SUMMARY:
This is an open-label phase 1 study to assess the safety, feasibility, pharmacokinetics and preliminary efficacy of autologous T cells co-expressing two CARs targeting the cryptic EGFR epitope 806 and IL3Ra2 (referred to as "CART-EGFR-IL13Ra2 cells"). Patients with newly diagnosed, EGFR-amplified, MGMT-unmethylated glioblastoma who have undergone maximal safe surgical resection will be approached for initial study participation. A two-step screening/eligibility process will be utilized. Following informed consent, subjects who meet Step #1 Eligibility Criteria will remain on study and complete a course of radiotherapy (60 Gy) without temozolomide as per their routine cancer care. If there is no overt evidence of disease recurrence/progression following radiotherapy, additional screening tests/procedures will be performed. Subjects who then meet Step #2 Eligibility Criteria will undergo apheresis collection to initiate cell product manufacturing and surgical placement of a CSF-Ventricular Reservoir to allow for intracerebroventricular injection of the CART-EGFR-IL13Ra2 cells. All subjects will receive a single fixed dose of CART-EGFR-IL13Ra2 cells on Day 0 via intracerebroventricular delivery.

ELIGIBILITY:
Step #1 Inclusion Criteria:

1. Signed informed consent form
2. Male or females age ≥ 18 years.
3. Patients with newly diagnosed, EGFR-amplified, MGMT-unmethylated glioblastoma (as defined by WHO 2021 Classification for CNS Tumors, including that the tumor must be IDH wildtype). The tumor must also have histopathologic evidence of glioblastoma (i.e., presence of microvascular proliferation and/or necrosis).
4. Patients must have undergone maximal safe resection of the tumor as per routine cancer care. Patients who have had a biopsy only are not eligible.
5. Tumor tissue positive for wild-type EGFR amplification by Neogenomics Laboratories
6. Karnofsky Performance Status ≥ 60%
7. Patient scheduled to receive 60 Gy of radiotherapy. Either photon or proton therapy is acceptable.

Step #1 Exclusion Criteria:

1. Active hepatitis B or hepatitis C infection
2. Class III/IV cardiovascular disability according to the New York Heart Association Classification.
3. Tumors with enhancing disease involving the thalamus, brain stem or spinal cord.
4. Tumors with an MGMT promoter methylation result of hypermethylated, methylated, low positive methylated, or indeterminate.
5. Multifocal disease if ≥ 1 focus of tumor has not undergone maximal safe resection
6. Severe, active co-morbidity that, in the opinion of the physician-investigator, would preclude participation in this study.
7. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
8. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10mg of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
9. Anticipated treatment plan that involves bevacizumab, any other systemic anti-neoplastic therapy, and/or tumor-treating fields as part of 1st line therapy.

Step #2 Inclusion Criteria:

1. Patient completed full course of radiotherapy to 60 Gy.
2. No overt evidence of disease recurrence/progression post-radiotherapy confirmed by RANO 2.0 criteria.
3. Karnofsky Performance Status ≥ 60%
4. Adequate organ function defined as:

   1. Serum creatinine ≤ 1.5x ULN or estimated creatinine clearance ≥ 30 mL/min and not on dialysis
   2. ALT/AST ≤ 3 x ILN
   3. Total bilirubin ≤ 2.0 mg/dl, except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome (≤ 3.0 mg/Dl)
   4. Left Ventricular Ejection Fraction (LVEF) ≥ 45% confirmed by ECHO/MUGA
   5. Must have minimum level of pulmonary reserve defined as > 92% on room air

Step #2 Exclusion Criteria:

1. Any active, uncontrolled infection.
2. Severe, active co-morbidity that, in the opinion of the physician-investigator, would preclude participation in this study.
3. Clinical or neurological decline related to disease and/or radiotherapy that, in the opinion of the physician-investigator, would preclude participation in this study.
4. Pregnant or nursing (lactating) patients. Participants of reproductive potential must agree to use acceptable birth control methods.
5. Receipt of prior bevacizumab therapy for their newly diagnosed glioblastoma.
6. Receipt of temozolomide for their newly diagnosed glioblastoma.
7. Anticipated post-radiotherapy maintenance treatment that includes tumor treating fields, bevacizumab, or any other anti-neoplastic therapies.
8. Enrollment in any other clinical trial for the treatment of their newly diagnosed glioblastoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2042-07 (Estimated); Study Completion 2042-07 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment related adverse events using NCI Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Type, frequency, severity, and attribution of adverse events
Occurrence of treatment-limiting toxicities (TLTs) | 28 days post-CAR T cell administration

SECONDARY OUTCOMES:
Proportion of enrolled subjects who receive study treatment as planned | 28 days following initial treatment with CART-EGFR-IL13Ra2 cells
  Evaluated based on the proportion of subjects who screen fail and those who receive any dose of CART-EGFR-IL13Ra2 cells.
Proportion of eligible subjects who receive study treatment as planned | 28 days following initial treatment with CART-EGFR-IL13Ra2 cells
Frequency of manufacturing failures | 3 months
  Proportion of subjects with CART-EGFR-IL13Ra2 products that fail to meet the product release criteria, out of the number of subjects in whom manufacturing was attempted.
  Proportion of subjects with CART-EGFR-IL13Ra2 products that fail to meet the assigned dose, out of the number of subjects in whom manufacturing was attempted.
Progression-free Survival (PFS) | Up to 15 years following CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria
Overall Survival (OS) | Up to 15 years following initial CART-EGFR-IL13Ra2 administration
  Time from initial study treatment to the date of death from any cause.
Objective Response Rate (ORR) | Up to 12 months following CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria (in subjects with measurable disease at the time of study treatment); Proportion of subjects with confirmed CR and PR.
Duration of response (DOR) | Up to 15 years following initial CART-EGFR-IL13Ra2 administration
  Per RANO 2.0 criteria (in subjects with measurable disease at the time of study treatment); Time from the date when a response of confirmed CR/PR is first met to the date of confirmed disease progression, death or receipt of alternative treatment other than CART-EGFR-IL13Ra2 retreatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bagley, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States